CLINICAL TRIAL: NCT02838160
Title: Effectiveness of Different Educational Strategies on the Knowledge, Attitude, and Practice ( KAP), Psychological and Clinical Outcomes in Intensive Care Unit: A Triple-blinded Randomized Controlled Follow-up Study
Brief Title: Effectiveness of Different Educational Strategies on the KAP, Psychological and Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Shahid Beheshti University (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Post doc, PhD, RN, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAP BMSU
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Ventilator-associated Pneumonia
Keywords: educational strategies; KAP; psychological and clinical outcomes; intensive care unit; follow-up study; RCT
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- booklet Group (Experimental)
  Interventions: Behavioral: Routine Care; Behavioral: Routine care Plus the designed booklet
- Oral presentations group (Experimental)
  Interventions: Behavioral: Routine Care; Behavioral: Routine care Plus the designed booklet; Behavioral: Routine care Plus the designed booklet Plus participation in oral presentations
- Clinical teaching in bedside Group (Experimental)
  Interventions: Behavioral: Routine Care; Behavioral: Routine care Plus the designed booklet; Behavioral: Routine care Plus the designed booklet Plus participation in oral presentations; Behavioral: Routine care Plus the designed booklet Plus participation in oral presentations Plus clinical teaching in bedside

INTERVENTIONS:
Behavioral: Routine Care — After baseline measurement, Group 1 did not receive any intervention or education.
Behavioral: Routine care Plus the designed booklet — Group 2 received only the designed booklet without any participation in the oral presentation.
Behavioral: Routine care Plus the designed booklet Plus participation in oral presentations — Group 3 participated in oral presentations 14 days after completing self-study booklet. Interactive, standardized and mandatory oral presentations were held five times to ensure maximum attendance of the three nursing shifts.
  Arms: Clinical teaching in bedside Group; Oral presentations group
Behavioral: Routine care Plus the designed booklet Plus participation in oral presentations Plus clinical teaching in bedside — The Group 4 received clinical teaching in bedside after completing self-study booklet and a series of interactive, standardized and mandatory 90-120-minute oral presentations.
  Arms: Clinical teaching in bedside Group

SUMMARY:
A randomized controlled triple blinded clinical trial with repeated measurements. The reporting of this study complies with the CONSORT (Consolidated Standards of Reporting Trials) statement for trials of non-pharmacological treatments.

The first aim of the study was to evaluate the effectiveness of the three competing interventions on the critical care nurses' knowledge of, attitudes toward and adherence to 17 ventilator bundle components; the second aim was to determine the effectiveness of adherence to 17 ventilator bundle components with pre-defined ventilator bundle on the psychological factors of critical care nurses including nurses' stressors in intensive care unit (ICU), perceived stress, trait and state anxieties; the third aim was to evaluate their impact on the clinical outcomes; and the fourth aim was comparing KAP and psychological factors with clinical outcomes.

DETAILED DESCRIPTION:
The multi-center study was conducted in four academic teaching hospitals in Tehran, Iran. The study consisted of a 3-month baseline observation period (October 2011-December 2011, Period 1), followed by a 6-month intervention period (January 2012 to June 2012) and a 3 (July 2012-September 2012, Period 2), 15 (October 2012-December 2013, Period 3) and 21-months (January 2014-June 2015, Period 4) follow-up periods. The protocol for Evidence based guidelines (EBGs) for preventing VAP remained unchanged throughout the study period in every ICU.

Consecutive adult patients (age ≥18 years) who were admitted to the mixed medical-surgical ICUs (>72 hours) and received invasive ventilation (>48 hours) were enrolled and monitored daily for the development of ventilator-associate pneumonia (VAP) until ICU discharge or death. Patients with any limitation of code status were excluded from the study. Convenience sample of critical care nurses were recruited through letters and telephone and face-to-face invitations. Inclusion criteria were holding a degree qualification as a registered nurse and being a direct care provider (bedside). Nurses with less than one year experience in critical care unit or working less than whole study period were excluded. An investigator at each participating medical center was responsible for initial screening and enrollment.

The sample size was determined through power analysis, which revealed that a sample size of 40 participants was required to detect a 20% difference between VAP rates in each group (α = 0.05, 1-β = 0.9; dropout = 20%). The estimation of the effect size based on a previous VAP surveillance, conducted from March 2010 to December 2010 (unpublished data).

Included nurses were randomly assigned to control or one of the three competing intervention group (allocation ratio of 1:4). Randomization was accomplished using Random Allocation Software© (RAS; Informer Technologies, Inc.). Block randomization was performed by a computer-generated randomization list prepared by blinded biostatistician who had no clinical involvement in the trial. All nurses, data collectors, and statistician were blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Holding a degree qualification as a registered nurse
* being a direct care provider (bedside)

Exclusion Criteria:

* Nurses with less than one year experience in critical care unit
* working less than whole study period were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
VAP Occurrence | One year
  VAP Occurrence according to the clinical sings and symptoms and laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Amir Vahedian-azimi, Postdoc, Principal Investigator — Baqiyatallah Universiy of Medical Sciences